CLINICAL TRIAL: NCT06966843
Title: Dantrolene in Statin-induced Myopathy
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Reem Alaa Abdel Samie, teacher assistant in Delta University for science and technology, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dan1199
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Statins Induced Myopathy
MeSH Terms: interventions — Dantrolene

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either dantrolene or placebo for 4 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dantrolene Group (Experimental): Participants will receive oral dantrolene 25 mg capsule once daily for 4 weeks. Dose may be increased to 50 mg daily based on tolerance and response. Dantrolene is used to evaluate its potential effect on muscle symptoms and biomarkers in statin-induced myopathy.
  Interventions: Drug: Dantrolene
- Placebo Group (Placebo Comparator): Participants will receive a matching oral placebo capsule once daily for 4 weeks, designed to mimic dantrolene in appearance. This arm serves as the control to assess the efficacy and safety of dantrolene in comparison to placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dantrolene — Dantrolene sodium capsule 25 mg orally once daily for 4 weeks. Dose may be titrated to 50 mg daily after 1 week if tolerated. Used to assess impact on muscle pain and biomarkers of muscle injury in patients with statin-induced myopathy.
  Other Names: Dantrium, Ryanodex
  Arms: Dantrolene Group
Drug: Placebo — Oral placebo capsule matching dantrolene in size and appearance, administered once daily for 4 weeks.
  Arms: Placebo Group

SUMMARY:
Statins are one of the most efficient drugs for the treatment of hypercholesterolemia which is considered as one of the main risk factors for atherosclerosis., and therefore they are frequently prescribed medications [1-2]. However, statins therapy is associated with myotoxicity. This effect of different severity ranges forms myopathy, myalgia, myositis, and rhabdomyolysis [3].

Different studies set a number of hypotheses to explain the pathophysiological events of statin-induced myopathy. These hypotheses include disturbance of mitochondrial function resulting in cytoplasmic Ca2+ overload as well as decreased level of the potent antioxidant and membrane stabilizer coenzyme Q10/ubiquinone [4-5] This study tries to introduce a complementary therapy that targets these molecular events. This therapeutic protocol includes dantrolene the muscle relaxant that acts as a ryanodine receptor (RYR) antagonist and thus decreases Ca release in cytoplasm.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-75 years Currently receiving statin therapy for at least 4 weeks Clinical symptoms suggestive of statin-induced myopathy (e.g., muscle pain, weakness) Elevated serum creatine kinase (CK) ≥1.5x upper limit of normal Able and willing to provide informed consent Willing to discontinue statins during the study period (if protocol requires)

Exclusion Criteria:

Known hypersensitivity to dantrolene History of severe liver disease or abnormal liver function tests (ALT or AST > 2x ULN) Use of interacting drugs that may increase dantrolene toxicity (e.g., calcium channel blockers like verapamil) Renal impairment (e.g., serum creatinine >2.0 mg/dL) Diagnosed neuromuscular disorders unrelated to statins (e.g., ALS, muscular dystrophy) Pregnant or breastfeeding women Participation in another clinical trial within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2027-10 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Change in Creatine Kinase (CK) Level | Baseline and 4 weeks after intervention start
  Evaluation of the effect of dantrolene on serum creatine kinase, a biomarker of muscle injury, in statin-induced myopathy.

SECONDARY OUTCOMES:
Change in Muscle Pain Score (Visual Analog Scale) | Baseline and Week 4
  Assessment of self-reported muscle pain severity using a 10-point VAS. Time Frame: Baseline and Week 4
Change in Serum Lactate Dehydrogenase (LDH) Level | Baseline and Week 4
  LDH as an additional marker of muscle damage.
Number of Participants With Adverse Effects Related to Dantrolene | Throughout the 4-week intervention period
  Safety evaluation of dantrolene use over the study period.